CLINICAL TRIAL: NCT02873806
Title: A Prospective Evaluation of Open-angle Glaucoma Subjects on Two Topical Hypotensive Medications (One a Prostaglandin) Treated With Two Trabecular Micro-bypass Stents (iStent Inject) and a Postoperative Topical Prostaglandin
Brief Title: Two Trabecular Micro-bypass Stents & Postoperative Travoprost to Treat Glaucoma Subjects on Two Hypotensive Agents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCF-039
Record Dates: First submitted 2016-08-11; First posted 2016-08-22 (Estimated); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Open-angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Travoprost; Tobramycin; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2 micro-bypass stents & travoprost (Other): Two iStent inject micro-bypass stents and topical travoprost
  Intervention:
  * Implantation of two iStent inject micro-bypass stents
  * Tobramycin
  * Dexamethasone
  Interventions: Procedure: Implantation of two iStent inject micro-bypass stents; Drug: Topical travoprost; Device: Two iStent inject micro-bypass stents; Drug: Tobramycin; Drug: Dexamethasone

INTERVENTIONS:
Procedure: Implantation of two iStent inject micro-bypass stents — - Implantation of two trabecular micro-bypass stents (iStent inject) in a standalone procedure (i.e., without cataract surgery).
  Other Names: iStent inject
Drug: Topical travoprost — - Topical travoprost (0.004%, 1 drop each evening in study eye) started on postoperative Day 1.
  Other Names: travoprost
Device: Two iStent inject micro-bypass stents — - Two trabecular micro-bypass stents (iStent inject) implanted in a standalone procedure.
  Other Names: iStent inject
Drug: Tobramycin — Topical antibiotic (tobramycin):
  1 drop four (4) times per day in the study eye for one week (in cases of allergy or contraindication, Polytrim (polymyxin B sulfate + trimethoprim sulfate ophthalmic solution, USP, or equivalent) may be used as an alternative medication) .
Drug: Dexamethasone — Topical anti-inflammatory medication (dexamethasone ophthalmic suspension 0.1%):
  * Week 1: 1 drop four (4) times per day in the study eye
  * Week 2: 1 drop three (3) times per day in the study eye
  * Week 3: 1 drop two (2) times per day in the study eye
  * Week 4: 1 drop one (1) time per day in the study eye

SUMMARY:
The study objective was to evaluate the intraocular pressure (IOP) lowering effect of two iStent devices in eyes of subjects with primary open-angle glaucoma, washed out of two anti-glaucoma medications (one a Prostaglandin) prior to stent implantation.

DETAILED DESCRIPTION:
The study design is as follows:

* Prospective, single-arm study.
* Subjects with open-angle glaucoma and medicated IOP > 18 mmHg and ≤ 30 mmHg.
* Subjects on two topical ocular hypotensive medications (one a prostaglandin).
* Implantation of two iStent inject devices (if IOP is < 6 mmHg, at any point during the postoperative follow-up, medication will not be prescribed or will be discontinued).
* IOP will be measured by two (2) observers to minimize bias; observer 1 will look through the slit lamp and turn the dial with readings being masked, and observer 2 will document the IOP.
* Follow-up through 60 months postoperative (or up to 61 months if subject needs to undergo terminal washout).
* Descriptive statistics will be tabulated.
* Medical therapy considered necessary for the subject's welfare can be implemented at any time during the study at the investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

Screening Exam Inclusion Criteria:

* Phakic patients or pseudophakic patients with posterior chamber intraocular lenses (PC-IOLs)
* Primary open-angle glaucoma (including pigmentary or pseudoexfoliative)
* C/D ratio ≤ 0.9
* Visual field defects, or nerve abnormality characteristic of glaucoma
* Two topical hypotensive medications at time of screening exam
* IOP > 18 mmHg and ≤ 30 mmHg (medicated) at screening exam
* Study eye BCVA 20/100 or better
* Normal angle anatomy as determined by gonioscopy
* Absence of peripheral anterior synechia (PAS), rubeosis or other angle abnormalities that could impair proper placement of stent

Baseline Exam Inclusion Criteria:

* Subject has completed appropriate medication washout
* Mean IOP > 22 mmHg and ≤ 38 mmHg after anti-glaucoma medication washout period
* A 3mmHg IOP increase over screening mean IOP

Exclusion Criteria:

Screening Exam Exclusion Criteria:

* Aphakic patients or pseudophakic patients with anterior chamber IOLs (AC-IOLs)
* Prior stent implantations (study eye)
* Traumatic, uveitic, neovascular, or angle-closure glaucoma; or glaucoma associated with vascular disorders
* Functionally significant visual field loss, including severe nerve fiber bundle defects
* Prior incisional glaucoma surgery
* Prior SLT within 90 days prior to screening
* Prior ALT
* Iridectomy or laser iridotomy
* Ineligibility for ocular hypotensive medication washout period as determined by the investigator.
* Any active corneal inflammation or edema (e.g., keratitis, keratoconjunctivitis, keratouveitis)
* Clinically significant corneal dystrophy (e.g., bullous keratopathy, Fuch's dystrophy); any guttata
* Corneal surgery (prior or anticipated) of any type (including LASIK, LASEK, PRK, etc.) that may interfere with IOP measurement reliability
* Corneal opacities that would inhibit visualization of the nasal angle
* Congenital or traumatic cataract
* Retinal or optic nerve disorders that are not associated with the existing glaucoma condition
* Elevated episcleral venous pressure such as associated with: active thyroid orbitopathy; cavernous sinus fistula; Sturge-Weber syndrome; orbital tumors; orbital congestive disease
* Clinically significant sequelae from trauma
* Chronic ocular inflammatory disease or presence of active ocular inflammation

Baseline Exam Exclusion Criteria:

* Subject did not complete medication washout
* Mean IOP < 22 mmHg or > 38 mmHg after anti-glaucoma medication washout
* Subject does not have a 3mmHg IOP increase over screening mean diurnal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2019-11-08 (Actual)

PRIMARY OUTCOMES:
Mean intraocular pressure reduction of 20% or more versus baseline with reduction of 1 medication | 12 months postoperative

SECONDARY OUTCOMES:
Mean intraocular pressure of 18 mmHg or less versus baseline with reduction of 1 medication | 12 months postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Lilit Voskanyan, MD, PhD, Principal Investigator — S.V. Malayan Eye Center
Locations (1):
- S.V. Malayan's Ophtalmology Centre, Yerevan, Armenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berdahl J, Voskanyan L, Myers JS, Hornbeak DM, Giamporcaro JE, Katz LJ, Samuelson TW. Implantation of two second-generation trabecular micro-bypass stents and topical travoprost in open-angle glaucoma not controlled on two preoperative medications: 18-month follow-up. Clin Exp Ophthalmol. 2017 Nov;45(8):797-802. doi: 10.1111/ceo.12958. Epub 2017 Jun 2. PMID 28384377